CLINICAL TRIAL: NCT04971824
Title: The Effect of Physiotherapy on Treatment Success by Assisted Reproductive Technologies
Brief Title: Physiotherapy in Assisted Reproductive Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klaudia Fabičovic, PT (Other)
Responsible Party: Sponsor-Investigator, Klaudia Fabičovic, PT, Master of Physiotherapy, Charles University, Czech Republic
Organization: Charles University, Czech Republic (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GA UK 184121
Record Dates: First submitted 2021-07-07; First posted 2021-07-22 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Infertility
Keywords: physiotherapy; assisted reproductive technologies; conception
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physiotherapeutic arm (Experimental): There will be the physiotherapeutic intervention, total duration for each participant is three months.
  The participants will be asked to fill three validated questionnaires in the beginning and in the end of study and keep records of their exercises, period and ovulation in their diaries.
  Interventions: Procedure: Physiotherapeutic intervention

INTERVENTIONS:
Procedure: Physiotherapeutic intervention — The physiotherapy consists in performing visceral manipulation of the pelvic and abdomen organs as well as doing special exercises (volunteers get a handout with instructions on how to exercise). The exercises include ones from the Mojzis´s method, Dynamic neuromuscular stabilisation, yoga or other therapeutic methods used by physiotherapists.

SUMMARY:
Research examines the effect of physiotherapy on treatment success by assisted reproductive technologies. It is based on a treatment of infertility by physiotherapeutic intervention after which the participants will undergo a treatment of assisted reproductive technologies (in vitro fertilisation). The work hypothesis is that physiotherapeutic treatment of female infertility improves the chances of conception by assisted reproductive technologies.

DETAILED DESCRIPTION:
This is an intervention study which also shows how physiotherapists can improve cooperation between two professionals (gynaecologists and physiotherapists). The study is based on physiotherapeutic intervention which consist of three months of physiotherapy.

The physical therapy program consists of 10 individual therapeutic sessions. Every session lasts 45 minutes, frequency of the first six sessions is once a week, frequency of the last four sessions is once every two weeks. The duration for each participant is three months.

The participants will be examined by the physiotherapist during first and last therapy session and they will be asked to fill questionnaires and to keep records of their exercises, period and ovulation in their diaries. There will be three validated questionnaires:

The 36-Item Short Form Health Survey, which measures a health-related quality of life, also the State-Trait Anxiety Inventory which measures state and trait anxiety and the last one is the Female Sexual Function Index which measures sexual function in women. The participants will be asked to do physiotherapeutic exercises as self-treatment every day according to a handout they get at the first therapy session.

The results from intervention group will be compared to control group in which we use retrospective data (from year 2019) from Centre of Assisted Reproduction of General University Hospital in Prague. We will compare the number of women treated by assisted reproductive technologies but without physiotherapeutic intervention.

To sum up, in this study we compare the number of women who conceived following the assisted reproductive technologies with and without physiotherapeutic intervention.

ELIGIBILITY:
Inclusion Criteria:

* nullipara
* age (18-39 years)
* in the past at minimum one failed attempt of conception by assisted reproductive technologies
* duration of infertility at minimum one year,
* Body Mass Index (BMI) 18,5-34,9 according to the World Health Organization

Exclusion Criteria:

* acute or chronic serious disease
* taking oral contraceptive pills for the last six months

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — The eligibility is based on gender because the study examines the effect of physiotherapy on woman who undergo treatment by assisted reproductive technologies.
Enrollment: 42 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2022-04-20 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
The effect of combination treatment of physiotherapy and assisted reproductive technologies | The total duration for each participant is three months.
  The number of woman who conceived after treatment consisted of physiotherapy and follow- up treatment by assisted reproductive technologies compared to the number of women who underwent treatment by assisted reproductive technologies without physiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Klaudia Fabičovic, Principal Investigator — First Faculty of Medicine, Charles University, General University Hospital in Prague, Department of Rehabilitation and Sports Medicine, Second Faculty of Medicine, Charles University and University Hospital Motol, Prague, Czech republic
Locations (1):
- First Faculty of Medicine, Charles University, General University Hospital in Prague, Department of Rehabilitation and Sports Medicine, Second Faculty of Medicine, Charles University and University Hospital Motol, Prague, Czech republic, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Yes
Some specific individual participant data will be shared (demographic data, the number of women who conceived in the end of study)
Supporting Information: CSR